CLINICAL TRIAL: NCT00677820
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of a Trivalent Vaccine of New 6:2 Influenza Virus Reassortants in Healthy Adults
Brief Title: A Prospective Study to Evaluate the Safety of a New Trivalent Intranasal Influenza Vaccine
Acronym: MI-MA182
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Raburn Mallory M.D.\Senior Director, Clinical Development, MedImmune LLC, an affiliate of AstraZeneca AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-MA182
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Influenza
Keywords: Influenza; FluMist; vaccine; prevention; trivalent
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trivalent influenza virus vaccine (Experimental): Frozen trivalent vaccine containing new strains
  Interventions: Biological: Trivalent influenza virus vaccine
- Placebo (Placebo Comparator): treatment with placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Trivalent influenza virus vaccine — Trivalent vaccine was supplied in intranasal sprayers containing a total volume of 0.5 ml of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10:7 FFU (fluorescent focus units) of each of three cold-adapted, attenuated, 6:2 reassortant influenza strains A/South Dakota/6/07 (H1N1), A/Uruguay/716/07 (H3N2), and B/Florida/4/2006.
  Arms: Trivalent influenza virus vaccine
Biological: Placebo — Placebo was supplied in intranasal sprayers containing 0.5 ml of sucrose-phosphate buffer.
  Arms: Placebo

SUMMARY:
This prospective annual release study was designed to assess the safety of a trivalent influenza virus vaccine using a new strain recommended for the 2008-2009 influenza season not previously contained in the trivalent intranasal FluMist vaccine. Three hundred healthy adults received a single dose of vaccine or placebo and were followed for 180 days.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind, placebo-controlled release study. Eligible subjects were randomly assigned in a 4:1 fashion to receive a single dose of trivalent vaccine or placebo by intranasal spray. Randomization was stratified by site. Each subject received 1 dose of study vaccine on Study Day 0. The duration of study participation for each subject was the time from study vaccination through 180 days after study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 49 years of age (not yet reached their 50th birthday) at the time of study vaccination
* Healthy by medical history and health assessment
* Sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral, implanted, injectable, or transdermal contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for at least 30 days prior to study vaccination, and must agree to continue using such precautions for at least 90 days after study vaccination; the subject must also have a negative serum or urine pregnancy test within 14 days prior to study vaccination (if screening and study vaccination do not occur on the same day) and on the day of study vaccination prior to randomization
* Sexually active males, unless surgically sterile, must use an effective method of birth control (condom or abstinence) and must agree to continue using such precautions for at least 30 days after study vaccination
* Available by telephone
* Provide written informed consent (and HIPAA authorization, if applicable)
* Ability to understand and comply with the requirements of the protocol, as judged by the investigator
* Ability to complete follow-up period of 180 days after study vaccination as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of the vaccine, including egg or egg protein
* History of hypersensitivity to gentamicin
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (eg, asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (>100.0°F oral or equivalent) and/or clinically significant respiratory illness (eg, cough or sore throat) within 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including HIV infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome
* A household contact who is severely immunocompromised (eg, hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual requires care in a protective environment); subject should additionally avoid close contact with severely immunocompromised individuals for at least 21 days after study vaccination
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 180 days after study vaccination (use of licensed agents for indications not listed in the package insert is permitted)
* Expected receipt of anti-pyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after study vaccination Note: A daily dose of up to 81 mg of aspirin for prophylactic use is not considered a contraindication to enrollment.
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after study vaccination
* Nursing mother
* Employee of the research center, any individual involved with the conduct of the study, or any family member of such individuals
* Any condition (eg, chronic cough, allergic rhinitis) that, in the opinion of the investigator, would interfere with evaluation of the vaccine or interpretation of study results

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Covance, Daytona Beach, Daytona Beach, Florida
  - Covance, Portland, Portland, Oregon
  - Covance, Austin, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 subjects were enrolled and randomized in the study between 09Jun2008 and 10Jun2008 at 3 sites in the USA.
Groups:
- Trivalent Influenza Virus Vaccine: Frozen trivalent vaccine containing the 3 new strains was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 fluorescent focus units (FFU) of each of 3 influenza virus strains type A/South Dakota/6/07 (H1N1), A/Uruguay/716/07 (H3N2), and B/Florida/4/2006. A single dose of investigational product was administered on Day 0.
- Placebo: Placebo was supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose-phosphate buffer and egg allantoic fluid. A single dose of investigational product was administered on Day 0.
Period: Overall Study
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Started | 240 | 60
Completed | 239 | 60
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo | Total
Number analyzed (Participants) | 240 | 60 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 31.2 (8.3) | 32.0 (9.3) | 31.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 43 | 194
  Male | 89 | 17 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 15 | 54
  Not Hispanic or Latino | 201 | 45 | 246
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 13 | 4 | 17
  White | 210 | 49 | 259
  More than one race | 4 | 2 | 6
  Other | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 240 | 60 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Fever
Description: Fever was defined as oral temperature greater than or equal to 101 degrees Fahrenheit.
Time Frame: Days 0-7
Population: Safety population Evaluable for Solicited Symptoms were subjects who received any study vaccine and experienced any follow-up for safety were considered evaluable for safety.
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants | 3 | 0

2. Secondary Outcome: Number of Subjects Reporting All Solicited Symptoms Post-treatment Days 0-7
Time Frame: Days 0-7
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 59
participants
  Any solicited symptom | 101 | 20
  Fever > 100F | 4 | 1
  Fever >= 101F | 3 | 0
  Fever > 102F | 0 | 0
  Fever > 103F | 0 | 0
  Runny nose | 52 | 6
  Sore throat | 32 | 7
  Cough | 7 | 2
  Vomiting | 2 | 0
  Muscle aches | 8 | 2
  Chills | 5 | 2
  Decreased activity | 20 | 5
  Headache | 41 | 8

3. Secondary Outcome: Number of Subjects Reporting Any Adverse Event (AE) Post-treatment
Time Frame: Days 0-7
Population: Subjects who received any study vaccine and experienced any follow-up for safety were considered evaluable for safety.
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants | 17 | 3

4. Secondary Outcome: Number of Subjects Reporting All Solicited Symptoms Post-treatment Days 0-14
Time Frame: Days 0-14
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 59
participants
  Any solicited symptom | 108 | 27
  Fever > 100F | 4 | 2
  Fever >= 101F | 3 | 0
  Fever > 102F | 0 | 0
  Fever > 103F | 0 | 0
  Runny nose | 58 | 7
  Sore throat | 37 | 8
  Cough | 10 | 4
  Vomiting | 3 | 1
  Muscle aches | 12 | 3
  Chills | 5 | 3
  Decreased activity | 24 | 5
  Headache | 44 | 14

5. Secondary Outcome: Number of Subjects Reporting Any AEs Post Treatment
Time Frame: Days 0-14
Population: Subjects who received any study vaccine and experienced any follow-up for safety were considered evaluable for safety.
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants | 20 | 5

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) and Significant New Medical Conditions (SNMC)
Description: SAEs were those that resulted in death; were life-threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a congenital anomaly/birth defect in the offspring of a study participant; or were an medical event that may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed above.
  An SNMC was a newly diagnosed medical condition of a chronic, ongoing nature and assessed by the investigator as medically significant.
Time Frame: Days 0-28
Population: Subjects who received any study vaccine and experienced any follow-up for safety were considered evaluable for safety.
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants
  Total subjects reporting > 1 SAE | 1 | 0
  Total subjects reporting > 1 SNMC | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting SAEs and SNMCs
Description: as for outcome 6
Time Frame: Days 0-180
Population: Subjects who received any study vaccine and experienced any follow-up for safety were considered evaluable for safety.
Measure: Number; unit: participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
participants
  Total subjects reporting > 1 SAE | 3 | 1
  Total subjects reporting > 1 SNMC | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms, AEs, and concomitant medication use were collected from administration of study vaccine through Study Day 14. Serious adverse events and SNMCs were collected from administration of study vaccine through Study Day 180.
Description: Adverse events and SAEs were graded by severity (mild, moderate, severe) and relationship to study vaccine (none, remote, possible, probable, definite).
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 3/240 | 1/60
Other Adverse Events (participants affected / at risk) | 12/240 | 5/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent Influenza Virus Vaccine (N=240) | Placebo (N=60)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent Influenza Virus Vaccine (N=240) | Placebo (N=60)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restricion is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.